CLINICAL TRIAL: NCT03708913
Title: Deep Brain Stimulation for Hypothalamic Obesity: A Surgical & Neuroimaging Study
Brief Title: Neuromodulation for Hypothalamic Obesity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants have been able to qualify for study
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Honey, Professor & Neurosurgeon, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H16-01595
Record Dates: First submitted 2016-12-08; First posted 2018-10-17 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Craniopharyngioma; Hypothalamic Obesity; Metabolic Syndrome
MeSH Terms: conditions — Craniopharyngioma; Sexual Infantilism; Metabolic Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-Label Lateral Hypothalamic DBS Stimulation (Experimental): Open-label lateral hypothalamic DBS stimulation for 1 year.
  Interventions: Device: Hypothalamic Deep Brain Stimulation

INTERVENTIONS:
Device: Hypothalamic Deep Brain Stimulation — One-year continuous hypothalamic deep brain stimulation

SUMMARY:
The balance between hunger and satiety is imperative for an individual's survival and overall health.). Without this balance, individuals can become morbidly obese or lack adequate nutrition for survival. Craniopharyngioma (CP) is a benign tumour that occurs at the base of the brain in children. Unfortunately, pediatric neurosurgeons sometimes inadvertently destroy a child's satiety centre during CP tumour removal surgery. This leaves the child with a post-operative complication: an insatiable appetite. This form of obesity is called "hypothalamic obesity". This study is designed to investigate Deep Brain Stimulation for hypothalamic obesity in n=6 young adults who have stabilized tumours.

DETAILED DESCRIPTION:
For young adults with destroyed satiety centres due to childhood CP surgery, we believe directly re-balancing the brain's control of hunger and satiety is necessary for sustained and long-term therapy. n=6 patients will be recruited in this Phase 1 DBS trial. The proposed research will hope to improve personal health among the young adults involved in this study by improving quality of life and avoiding long-term cardiovascular morbidities. Furthermore, this study will elucidate what brain regions drive excessive hunger and develop a treatment that attempts to reverse these abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hypothalamic obesity following craniopharyngioma tumour removal
* Treatment refractory to pharmacological interventions such as growth hormone therapy and anti-obesity medications

Exclusion Criteria:

* Unable to give consent or unmanaged psychiatric condition

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events That Are Related to surgery and Post-Operative Side Effects | 12 months

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 12 months
  Measuring BMI(kg/m^2) following 12 months of constant stimulation
Hyperphagia Questionnaire | 12 months
  Completion of hyperphagia questionnaire
SF-36 Quality of Life Questionnaire | 12 months
  Completion of QoL Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Leslie and Gordon Diamond Health Center, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Lustig RH. Hypothalamic obesity after craniopharyngioma: mechanisms, diagnosis, and treatment. Front Endocrinol (Lausanne). 2011 Nov 3;2:60. doi: 10.3389/fendo.2011.00060. eCollection 2011. PMID 22654817
- [Background] Lustig RH. Hypothalamic obesity: causes, consequences, treatment. Pediatr Endocrinol Rev. 2008 Dec;6(2):220-7. PMID 19202508
- [Background] Lustig RH, Post SR, Srivannaboon K, Rose SR, Danish RK, Burghen GA, Xiong X, Wu S, Merchant TE. Risk factors for the development of obesity in children surviving brain tumors. J Clin Endocrinol Metab. 2003 Feb;88(2):611-6. doi: 10.1210/jc.2002-021180. PMID 12574189
- [Background] Lustig RH, Rose SR, Burghen GA, Velasquez-Mieyer P, Broome DC, Smith K, Li H, Hudson MM, Heideman RL, Kun LE. Hypothalamic obesity caused by cranial insult in children: altered glucose and insulin dynamics and reversal by a somatostatin agonist. J Pediatr. 1999 Aug;135(2 Pt 1):162-8. doi: 10.1016/s0022-3476(99)70017-x. PMID 10431109
- [Background] Ho AL, Sussman ES, Zhang M, Pendharkar AV, Azagury DE, Bohon C, Halpern CH. Deep Brain Stimulation for Obesity. Cureus. 2015 Mar 25;7(3):e259. doi: 10.7759/cureus.259. eCollection 2015 Mar. PMID 26180683